CLINICAL TRIAL: NCT03840239
Title: Total Neoadjuvant trEatment to Increase the Clinical Complete reSponse Rate for diStal Locally Advanced Rectal Cancer (TESS)
Brief Title: TNT to Increase the Clinical Complete Response Rate for Distal LARC
Acronym: TESS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, WeiWei Xiao, Associate professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-FXY-149; 5010-2018-04 (Other: Sun Yat-sen University Cancer Center)
Record Dates: First submitted 2019-01-28; First posted 2019-02-15 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Rectal Cancer; Rectal Cancer Stage II; Rectal Cancer Stage III; Chemoradiation
Keywords: rectal cancer; chemoradiation; total neoadjuvant treatment
MeSH Terms: conditions — Rectal Neoplasms | interventions — XELOX; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TNT arm (Experimental): Drug: Neoadjuvant chemotherapy Capeox (Capecitabine + Oxaliplatin), 6 cycles; adjuvant chemotherapy, Capecitabine, 2 cycles or physicians' decision.
  External beam radiotherapy: Neoadjuvant, 50 Gy, 2 Gy/session; 25 fractions. Procedure: 'Watch and wait strategy' or surgery including local excision, intersphincter resection or total mesorectal excision or other kinds of surgeries.
  Interventions: Drug: Capecitabine, Oxaliplatin; Radiation: External beam radiotherapy; Procedure: Surgery; Other: Watch and wait strategy

INTERVENTIONS:
Drug: Capecitabine, Oxaliplatin — Drug: Capecitabine, Oxaliplatin
Radiation: External beam radiotherapy — External beam radiotherapy to the primary tumor, regional lymph nodes and clinical target volume
Procedure: Surgery — 'Local excision' or 'Intersphincter resection' or 'Total mesorectal excision' or other surgeries
Other: Watch and wait strategy — Watch and wait strategy recommendation and discussion for cCR patients

SUMMARY:
This is a open-label, single-arm study to investigate the safety and efficacy of total neoadjuvant treatment (TNT) in patients with locally advanced resectable rectal cancer.

DETAILED DESCRIPTION:
Standard treatment of rectal cancer is neoadjuvant capecitabine chemotherapy with radiotherapy, followed by total mesorectal excision.

A new concept suggests organ preservation as an alternative to rectal excision in good responders after neoadjuvant radiochemotherapy to decrease surgical morbidity and increase quality of life.

The rational is the fact that 15%-20% of patients have sterilized tumours after chemoradiotherpay for locally advanced rectal cancer. As compared to capecitabine alone, oxaliplatin and more intensified chemotherapy have been shown to increase tumor regression in the neoadjuvant chemoradiation setting. Meanwhile, prolong of time interval from the end of radiotherapy to assessment of tumor response could further increase pathologic complete response rate and complete clinical response rate.

The objective of this trial is to increase the rate of clinical complete response for distal rectal cancer patients by optimizing tumour response. The investigators expect to increase chance of clinical complete response by using total neoadjuvant treatment regimen as compared to conventional chemoradiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Rectal adenocarcinoma
* cT3-4aNany or cTanyN+
* Location ≤5 cm from the anal verge
* No distant metastasis
* No gastrointestinal obstruction or relieved obstruction
* No previous surgery of the rectum, no previous chemotherapy, no previous pelvic radiation, no previous biotherapy
* ECOG 0-1
* Expected survival length ≥ 2 years
* Age 18-70
* Sufficient bone marrow, kidney and liver function
* Effective contraception during the study
* Patient and doctor have signed informed consent

Exclusion Criteria:

* Distant metastasis
* Chronic intestinal inflammation and/or bowel obstruction
* Contra indication for chemotherapy and/or radiotherapy
* Previous pelvic radiotherapy or chemotherapy
* Severe renal, hepatic insufficiency (serum creatinine<30ml/min)
* Peripheral neuropathy > grade 1
* Pregnant or breast-feeding woman
* Certain or suspicious allergy to research drug
* Cachexia, organ dysfunction
* Active severe infection
* Multiple primary cancers
* Epileptic seizures
* Malignant history within 5 years, except cervical carcinoma in situ or cutaneous basal cell carcinoma
* Severe arrhythmia, cardiac dysfunction (NYHA grade III or IV )
* Uncontollable severe hypertesion
* Persons deprived of liberty or under guardianship
* Impossibility for compliance to follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2018-12-25 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical complete response | 1.5 year after diagnosis
  Rate of clinical complete response

SECONDARY OUTCOMES:
Ratio of sphincter preservation strategy | 1.5 year after diagnosis
  Number of patients with sphincter preservation through Watch and wait strategy, or local excision, or intersphincter resection, or low anterior resection, etc.
Rate of pathological complete response and tumor regression grade distribution | 1.5 year after diagnosis
  Rate of pathological complete response and tumor regression grade distribution
Acute toxicity | Within the first course of anti-tumor treatment
  Acute toxicity according to CTCAE 5.0
Rate of surgical complications | 1.5 year after diagnosis
  Rate of surgical complications
Long-term anal function | 1.5 year after diagnosis
  Long-term anal function according to Wexner Continence Grading Scale
Long-term toxicity grading | 3 year after the end of the first course of anti-tumor treatment
  Long-term toxicity grading according to CTCAE 5.0
ECOG standard score | 1.5 year after diagnosis
  ECOG standard score
3 year disease free survival | 3 year after the end of the first course of anti-tumor treatment
  3 year disease free survival
5 year overall survival | 5 year after the end of the first course of anti-tumor treatment
  5 year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: WeiWei Xiao, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided